CLINICAL TRIAL: NCT05031481
Title: National, Multicenter, Randomized, Double-blind, Phase II Clinical Trial to Evaluate the Efficacy and Safety of Different Doses of Venus Association in Patients With Vulvovaginal Candidiasis
Brief Title: Efficacy and Safety of Different Doses of Venus Association in Patients With Vulvovaginal Candidiasis.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS1819 - VENUS
Record Dates: First submitted 2021-08-26; First posted 2021-09-02 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Vulvovaginal Candidiasis
Keywords: Vulvovaginal Candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — butoconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VENUS 20 + 0,064 (Experimental): Venus association vaginal cream, single dose.
  Interventions: Drug: Venus 20 + 0,064
- VENUS 20 + 1 (Experimental): Venus association vaginal cream, single dose.
  Interventions: Drug: Venus 20 + 1
- VENUS 20 + 4 (Experimental): Venus association vaginal cream, single dose.
  Interventions: Drug: Venus 20 + 4
- Butoconazole nitrate 100 mg (Active Comparator): Butoconazole nitrate vaginal cream, single-dose containing 100 mg.
  Interventions: Drug: Butoconazole nitrate

INTERVENTIONS:
Drug: Venus 20 + 0,064 — Venus vaginal cream 20 + 0,064, single-dose.
  Arms: VENUS 20 + 0,064
Drug: Venus 20 + 1 — Venus vaginal cream 20 + 1, single-dose.
  Arms: VENUS 20 + 1
Drug: Venus 20 + 4 — Venus vaginal cream 20 + 4, single-dose.
  Arms: VENUS 20 + 4
Drug: Butoconazole nitrate — Butoconazole nitrate vaginal cream, 100 mg single-dose.
  Arms: Butoconazole nitrate 100 mg

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of different doses of Venus association in the treatment of vulvovaginal candidiasis.

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the informed consent forms;
* Age greater than or equal to 18 years;
* Female participants, post-menarche;
* Clinical diagnosis of vulvovaginal candidiasis, defined as white, fluid or creamy vaginal discharge, in addition to the following findings:
* Itching and one or more of the following signs and symptoms characterized as moderate or severe: vulvar/vaginal erythema, edema, burning, irritation, and excoriation;
* Normal vaginal pH;
* Preparation of KOH or saline from a sample taken from inflamed vaginal mucosa or secretions revealing yeast forms (hyphae or pseudohyphae) or growing yeast.

Exclusion Criteria:

* Any clinical and laboratory findings that, in the judgment of the investigator, may interfere with the safety of research participants;
* Participation in a clinical trial in the year prior to this study;
* Pregnancy or risk of pregnancy and lactating patients;
* Known hypersensitivity to any of the formula compounds;
* Virgin participants;
* Postmenopausal participants or with vaginal atrophy;
* Participants with other vaginal infections;
* Participants with recurrent vulvovaginal candidiasis;
* Participants using immunosuppressive drugs;
* Participants diagnosed with serious systemic diseases.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Time to first relief of symptoms | 0-24 hours
  Time to obtain moderate relief of at least one of the evaluated symptoms (itching, irritation or burning) after the application of the medication.

SECONDARY OUTCOMES:
Adverse events | 28 days
  Incidence and severity of adverse events recorded during the study.